CLINICAL TRIAL: NCT01580267
Title: Hepcidin and Anemia in Trauma
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lena Napolitano, MD, Principal Investigator, University of Michigan
Other Study IDs: HUM00053750
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Anemia
Keywords: Anemia in trauma
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Anemia (decreased number of red blood cells) is common in critically ill trauma patients admitted to an Intensive Care Unit and is associated with a high rate of blood transfusions. This "anemia of inflammation" is a result of three mechanisms: impaired iron regulation, shortened red blood cell life span, and reduced rate of erythropoiesis (a protein that helps make new red blood cells).

Hepcidin, a protein made in the liver, regulates iron and is decreased when iron in the blood is low. This can lead to anemia.

This research study is being conducted to learn how inflammation, hepcidin, and erythropoietin interact in critically ill patients. The findings will help in determining effective treatment for patients with anemia of inflammation.

DETAILED DESCRIPTION:
Anemia is common in trauma patients and is associated with a high rate of blood transfusion. The pathophysiology of this anemia is "anemia of inflammation" and develops via 3 mechanisms: impaired iron regulation, shortened red blood cell life span, and reduced rate of erythropoiesis. Once iron enters cells (enterocytes and macrophages), the iron export protein ferroportin controls egress. Hepcidin, a peptide made in the liver, is the key regulator of iron homeostasis. Hepcidin binds to ferroportin, leading to its ultimate degradation. Hepcidin reduces iron availability via 2 mechanisms: decreased absorption of iron across the GI tract and decreased release of iron from the reticuloendothelial system. It therefore induces a functional iron deficiency by shuttling iron into the macrophages and making it unavailable for erythropoiesis. Hepcidin is decreased by iron deficiency, most anemias, and tissue hypoxia. Hepcidin is upregulated by iron excess and inflammation. Hepcidin likely plays an important role in the acute inflammatory response that occurs with trauma. However, no studies have measured hepcidin in critically ill trauma patients. If serum hepcidin levels are elevated in trauma, this will confirm that inability to use existing iron stores is part of, if not key to, the anemia of trauma and critical illness. This has important implications since the use of blood transfusion for anemia treatment may further induce an inflammatory response with resultant suppression of native erythropoiesis.

The investigators hypothesize that hepcidin will be increased and erythropoietin decreased early after trauma and that resolution of anemia will not occur until late (28-31 days). By measuring time-dependent changes in hemoglobin, hepcidin, cytokine, and erythropoietin concentrations in trauma patients, the investigators can critically examine the inter-relationships to target potential therapeutic strategies for the treatment and amelioration of anemia in trauma and critical care.

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patient
2. Age 18 years or older
3. Admitted to ICU
4. Anemic (Hct < 34.5%)

Exclusion Criteria:

1. Pre-existing hematological disorder
2. Pre-existing diagnosis of anemia or other known iron disorder
3. Chronic renal failure
4. Use of recombinant erythropoietin
5. Treatment with systemic immunosuppressant or cytotoxic drugs
6. Pregnancy
7. Patients not expected to survive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients, 18 years of age or older, admitted to a University of Michigan ICU
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena M Napolitano, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States